CLINICAL TRIAL: NCT04313517
Title: Yoga@Work Intervention to Reduce Work Related Stress Among Information Technology Workers: Waitlist Controlled Trial
Brief Title: Yoga@Work Intervention to Reduce Work-related Stress Among Information Technology Workers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarogyam UK (Other)
Collaborators: Brunel University (Other); NMP Medical Research Institute (Other); Ananda Yoga (Hong Kong) (Unknown); Vrije Universiteit Brussel (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AUI01
Record Dates: First submitted 2020-03-17; First posted 2020-03-18 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Occupational Stress; Psychological Stress
MeSH Terms: conditions — Occupational Stress; Stress, Psychological | interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga@Work (Experimental): Yoga session were developed to practice at work anytime feasible.
  Interventions: Other: Yoga
- Wait list Control group (No Intervention): Control group with no intervention. After Intervention period, group was offered same sessions.

INTERVENTIONS:
Other: Yoga — Each yoga session included warm-up practices (for the large joints, spine, and extremities), Simple postures (Asana), breathing exercises (pranayama) and meditation/relaxation. All the yoga participants were given handouts to practice everyday at work as its feasible
  Arms: Yoga@Work

SUMMARY:
Over the last several decades, occupational stress at workplace comprise a major burden. Office based work are more prone to sedentary lifestyle, postural issues, workplace stress, repetitive strain injury, poor employee health. Workplace wellness programs has been very feasible access to employees at their own convenience and need. Yoga@Work Program was developed to suit the need for information technology workers.

ELIGIBILITY:
Inclusion Criteria:

* Information Technology employee, or trainee willing and able to participate in a 6-week self-care program during the work day.
* Willing to give informed consent

Exclusion Criteria:

* medical or psychiatric conditions limiting practice of yoga in general
* Cognitive impairment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2019-01-12 (Actual); Primary Completion 2019-06-18 (Actual); Study Completion 2019-09-21 (Actual)

PRIMARY OUTCOMES:
Reductions in occupational stress | From baseline to 6-week post intervention
  Perceived Stress Scale

SECONDARY OUTCOMES:
Mental health problems | From baseline to 6-week post intervention
  General Health questionnaires consists of 12 items, each assessing the severity of a mental problem

CONTACTS AND LOCATIONS:
Overall Officials: Neha Sharma, PhD, Principal Investigator — Aarogyam UK; Jaydeep Joshi, BAMS, Study Director — Aarogyam UK; Monomita Nandy, Study Chair — Brunel University
Locations (4):
- UNRI, Brussels, Belgium
- Ananda Yoga, Hong Kong, Hong Kong
- NMP Medical Research Institute, Jaipur, Rajasthan, India
- Yog-Kulam, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided